CLINICAL TRIAL: NCT01950247
Title: Evaluate the Utility of Serum Hepcidin Levels to Predict Response to Oral or IV Iron and Compare the Safety, Effect on QOL and Resource Utilization, of Injectafer® vs. IV Iron Standard of Care for the Treatment of IDA in an Infusion Center
Brief Title: Evaluate the Utility of Serum Hepcidin Levels to Predict Response to Oral or IV Iron
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT13032
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-11

CONDITIONS: Iron Deficiency Anemia (IDA)
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Injectafer (Experimental): 2 doses at 15 mg/kg for a maximum single dose of 750 mg given 7 days apart for a total of up to 1500 mg.
  Interventions: Drug: Injectafer
- IV Iron Standard of Care (SOC) (Active Comparator): At a dose and administration regimen as determined by the study site investigator
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: Injectafer — 2 doses at 15 mg/kg for a maximum single dose of 750 mg given 7 days apart for a total of up to 1500 mg.
  Other Names: Ferric Carboxymaltose (FCM)
  Arms: Injectafer
Drug: SOC
  Other Names: IV Iron Standard of Care
  Arms: IV Iron Standard of Care (SOC)

SUMMARY:
The main objective of this study is to compare the safety, effect on quality of life, and resource utilization of Injectafer vs. intravenous (IV) iron standard of care (SOC) for the treatment of iron deficiency anemia (IDA) in an infusion center setting. The study will also assess the ability of baseline serum hepcidin levels to predict if subjects will have a clinically meaningful hemoglobin response to oral iron therapy or to IV iron therapy.

DETAILED DESCRIPTION:
The main objective of this study is to compare the safety, effect on quality of life, and resource utilization of Injectafer vs. intravenous (IV) iron standard of care (SOC) for the treatment of iron deficiency anemia (IDA) in an infusion center setting. The study will also assess the ability of baseline serum hepcidin levels to predict if subjects will have a clinically meaningful hemoglobin response to oral iron therapy for 28 days or to IV iron therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age and able to give informed consent.
* Iron deficiency is the primary etiology of anemia.
* If using erythropoiesis stimulating agent (ESA), the subject must be using a dose consistent with package insert that has been stable for at least 30 days.
* Doses of potential myelosuppressive medications have been stable for at least 30 days.
* Females at risk of pregnancy must agree to use an acceptable form of birth control and have a negative serum or urine pregnancy test on the first day of dosing.

Exclusion Criteria:

* Hypersensitivity reaction to any component of Injectafer.
* Requires dialysis for treatment of chronic kidney disease (CKD).
* No evidence of iron deficiency.
* During the 10 day period prior to screening has been treated with intravenous iron.
* During the 30 day period prior to screening has been treated with a red red blood cell transfusion.
* Any non-viral infection.
* Known positive hepatitis with evidence of active disease.
* Received an investigational drug within 30 days of screening.
* Alcohol or drug abuse within the past 6 months.
* Hemochromatosis or other iron storage disorders.
* Estimated life expectancy of less than 6 months, or for cancer patients, an Eastern Cooperative Oncology Group (ECOG) Performance Status greater than 1.
* Pregnant or actively trying to become pregnant (a definitive negative result on a serum or urine pregnancy test performed on the first day of dosing will be required for study enrollment by any women of childbearing potential).
* Any other laboratory abnormality, medical condition or psychiatric disorders which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1025 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — American Regent, Inc.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Iron Standard of Care (SOC): At a dose and administration regimen as determined by the study site investigator
  Standard of Care (SOC)
Period: Overall Study
Arm/Group | IV Iron Standard of Care (SOC) | Injectafer
Started | 512 | 513
Completed | 455 | 467
Not Completed | 57 | 46
Not completed — Withdrawal by Subject | 28 | 13
Not completed — Lost to Follow-up | 18 | 16
Not completed — Physician Decision | 3 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Death | 1 | 1
Not completed — Not Defined | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- IV Iron Standard of Care (SOC): At a dose and administration regimen as determined by the study site investigator
  SOC
- Total: Total of all reporting groups
Arm/Group | Injectafer | IV Iron Standard of Care (SOC) | Total
Number analyzed (Participants) | 513 | 512 | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (16.58) | 55.7 (16.68) | 56.5 (16.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 421 | 409 | 830
  Male | 92 | 103 | 195
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 513 | 512 | 1025

OUTCOME MEASURES:

1. Primary Outcome: Multidimensional Assessment of Fatigue (MAF) Scores
Description: The MAF scale has 16 items that measure the Global Fatigue Index (GFI), a composite score of Items 1 through 15. Items 1 through 14 were measured on a scale of 1 to 10, with 1 = not at all and 10 = a great deal. Items 15 and 16 had categorical responses: degree of agreement from 0 to 4, with 0=no days and 4=every day. Then, a Global Fatigue Index (GFI) is calculated by summing specific items and averaging others. The final GFI score ranges from 1 (no fatigue) to 50 (severe fatigue). The resulting score is given as the mean value.
Time Frame: Baseline to Day 30
Population: Change from baseline to Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | IV Iron Standard of Care (SOC)
Number analyzed (Participants) | 264 | 269
units on a scale | -8.8 (11.38) | -8.1 (11.28)

2. Primary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI) Scores
Description: The WPAI consisted of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working using a scale of 0 to 10, with 0 = PROBLEM had no effect on my work and 10 = PROBLEM completely prevented me from working; 6 = degree health affected productivity in regular unpaid activities using a scale of 0 to 10, with 0 = PROBLEM had no effect on my daily activities and 10 = PROBLEM completely prevented me from doing my daily activities. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline and Day 30
Population: Change from baseline to Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | IV Iron Standard of Care (SOC)
Number analyzed (Participants) | 513 | 512
units on a scale
  Percent activity impairment due to problem: number analyzed (Participants) | 446 | 432
  Percent activity impairment due to problem | -15.2 (29.85) | -11.5 (29.43)
  Percent impairment while working due to problem: number analyzed (Participants) | 142 | 154
  Percent impairment while working due to problem | -13.2 (28.75) | -8.5 (24.44)
  Percent overall work impairment due to problem: number analyzed (Participants) | 142 | 154
  Percent overall work impairment due to problem | -13.4 (31.66) | -8.5 (25.89)
  Percent work time missed due to problem: number analyzed (Participants) | 149 | 156
  Percent work time missed due to problem | -3.2 (23.76) | -2.5 (17.23)

3. Primary Outcome: Treatment Satisfaction Questionnaire for Medication Version 1.4 Scores
Description: Participants rated 14 items with 4 domains. Scores for item 1 to 3, 9 to 11 and 14 ranged from 1=extremely dissatisfied to 7=extremely satisfied. Items 5 to 8, 12, 13 ranged from 1=extremely dissatisfied to 5=not at all dissatisfied. Item 4 was scored as: 0=No, 1=Yes. Effectiveness measured as ([{sum of item 1 to 3} - 3]/18)*100; if 1 question (Q) was missing: ([{sum of item 1 to 3} -2]/12)*100. Side-effect measured as if item 4=No, score=100; if not then ([{sum of item 5 to 8} -4]/16)*100; if 1 Q was missing: ([{sum of item 5 to 8} -3]/12)*100. Convenience measured as ([{sum of item 9 to 11} -3]/18)*100; if 1 Q was missing: ([{sum of item 9 to 11} - 2]/12)*100. Global satisfaction as ([{sum of item 12 to 14} -3]/14)*100; if item 12 or 13 was missing: ([{sum of item 12 to 14} -2]/10)*100; if item 14 was missing: ([{sum of item 12 and 13} -2]/8)*100. All domains had scale of 0 (no satisfaction) to 100 (best level of satisfaction), higher score equals greater satisfaction
Time Frame: Baseline and Day 30
Population: Change from baseline to Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | IV Iron Standard of Care (SOC)
Number analyzed (Participants) | 513 | 512
units on a scale
  Overall Satisfaction: number analyzed (Participants) | 456 | 438
  Overall Satisfaction | 72.6 (25.03) | 72.7 (21.07)
  Effectiveness: number analyzed (Participants) | 456 | 440
  Effectiveness | 69.3 (22.38) | 66.5 (21.75)
  Side Effects: number analyzed (Participants) | 95 | 102
  Side Effects | 63.5 (27.21) | 69.2 (21.00)
  Convenience: number analyzed (Participants) | 454 | 437
  Convenience | 78.9 (17.31) | 72.8 (20.00)

4. Primary Outcome: Short Form Health Survey, 12-Item (SF-12) v2 Quality of Life Scores.
Description: The SF-12 is a multipurpose short form to measure health status. There are 10 domains: Physical Composite Index (score range from 0-100); Physical Functioning Index (score range from 0-100); Role Limitation Physical Index (score range 0-100); Pain Index Score (score range from 0-100); General Health Index (score range from 0-100); Mental Health Composite Index (score range from 1-100); Vitality Index (score range from 0-100); Social Functioning Index (score rang 0-100); Role Limitation Emotional Index (score range 0-100); and SF-12 Mental Health Index (score range from 0-100), the higher the score means a better outcome. The overall scale and sub-scales were calculated with the standard SF-12 formulas.
Time Frame: Baseline and Day 30
Population: Change from Baseline to Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectafer | IV Iron Standard of Care (SOC)
Number analyzed (Participants) | 513 | 512
units on a scale
  Pain: number analyzed (Participants) | 458 | 438
  Pain | 1.6 (10.03) | 2.5 (10.52)
  Overall Physical Health Score: number analyzed (Participants) | 443 | 428
  Overall Physical Health Score | 3.3 (7.94) | 3.1 (8.33)
  Overall Mental Health Score: number analyzed (Participants) | 443 | 428
  Overall Mental Health Score | 3.7 (10.31) | 3.7 (10.39)
  Physical Functioning: number analyzed (Participants) | 457 | 437
  Physical Functioning | 3.6 (10.42) | 3.4 (10.45)
  Role Limitation Physical: number analyzed (Participants) | 458 | 436
  Role Limitation Physical | 4.0 (9.53) | 3.9 (9.25)
  General Health: number analyzed (Participants) | 457 | 439
  General Health | 3.2 (9.86) | 2.5 (9.84)
  Vitality: number analyzed (Participants) | 453 | 436
  Vitality | 7.7 (11.36) | 7.0 (11.53)
  Social Functioning: number analyzed (Participants) | 454 | 438
  Social Functioning | 3.6 (12.19) | 3.0 (11.47)
  Role Limitation Emotion: number analyzed (Participants) | 456 | 432
  Role Limitation Emotion | 2.7 (12.69) | 2.8 (12.62)
  Mental Health: number analyzed (Participants) | 452 | 436
  Mental Health | 2.9 (10.10) | 3.3 (9.62)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 30
Description: Adverse events were collected by systematic assessment
Arm/Group | Injectafer | IV Iron Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 1/513 | 1/512
Serious Adverse Events (participants affected / at risk) | 4/513 | 1/512
Other Adverse Events (participants affected / at risk) | 28/513 | 21/512
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=513) | IV Iron Standard of Care (SOC) (N=512)
Cardiac disorders (Cardiac disorders) | 4 (506) | 1 (486)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectafer (N=513) | IV Iron Standard of Care (SOC) (N=512)
Nausea (Gastrointestinal disorders) | 28 (506) | 21 (486)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes